CLINICAL TRIAL: NCT00797342
Title: A Phase 1, Randomized, Double Blind (Sponsor Open), Placebo Controlled, Single-Dose Escalation Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effect of PF-04629991 in Healthy Volunteers
Brief Title: A Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PF-04629991 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: B0881001
Record Dates: First submitted 2008-11-19; First posted 2008-11-25 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Healthy Volunteers
Keywords: rheumatoid arthritis First in human safety pharmacokinetics pharmacodynamics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- first of three dosing cohorts (Other)
  Interventions: Drug: PF-04629991
- second of three dosing cohorts (Other)
  Interventions: Drug: PF-04629991
- third of three dosing cohorts (Other)
  Interventions: Drug: PF-04629991

INTERVENTIONS:
Drug: PF-04629991 — Oral; Sequential single dose escalation; three fourteen-day treatment periods per subject in the first cohort; randomized sequence of treatments (one placebo and two PF-04629991 doses)
  Arms: first of three dosing cohorts
Drug: PF-04629991 — Oral; Sequential single dose escalation; three fourteen-day treatment periods per subject in the second cohort; randomized sequence of treatments (one placebo and two PF-04629991 doses)
  Arms: second of three dosing cohorts
Drug: PF-04629991 — Oral; sequential single dose escalation; three fourteen-day treatment periods per subject in the third cohort; randomized assignment to treatment (placebo or PF-04629991)
  Arms: third of three dosing cohorts

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of PF-04629991 in healthy subjects. Dose exploration will proceed in a step-wise manner, beginning with low doses not expected to have significant biological effects and proceeding to doses approximating or exceeding the anticipated therapeutic level. Doses to be explored may be limited by tolerability, and will not exceed levels previously shown to be tolerable in animals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking men and women
* body mass index 18-30 kg/m2

Exclusion Criteria:

* Women must not be able to have children
* no current infections

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics e.g., maximum concentration and area under the concentration-time curve | 2 weeks
Safety/Tolerability e.g., reported adverse events and safety laboratory studies | 2 weeks
Pharmacodynamics e.g., changes in a peripheral blood biomarker | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0881001&StudyName=A%20Study%20of%20the%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%20and%20Pharmacodynamics%20of%20PF-04629991%20in%20Healthy%20Volunteers